CLINICAL TRIAL: NCT05902195
Title: Improving Work Ability of Young Adults With Stroke Through Personal Resource Building and Inclusive Volunteering: A Randomised Controlled Trial
Brief Title: Improving Work Ability of Young Adults With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne HS Lo, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PVI
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Return to work
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A 2-arm, assessor-blind, randomised controlled trial will be conducted.
Who Masked: Outcomes Assessor
Masking Description: Assessor-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal Resource Building and Inclusive Volunteering Intervention (PVI) (Experimental): All participants in the intervention group will receive the intervention (PVI) in addition to usual care. PVI is a 6-week virtual programme aimed at building up young stroke survivors' personal resources for work through engaging in inclusive volunteering activities.
  Interventions: Behavioral: Personal Resource Building and Inclusive Volunteering Intervention (PVI)
- Control (Active Comparator): All participants in the control group will receive usual stroke care services such as medical or health services offered by the hospitals or community-based organisations.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Personal Resource Building and Inclusive Volunteering Intervention (PVI) — PVI is a 6-week virtual programme aimed at building up young stroke survivors' personal resources for work through engaging in inclusive volunteering activities.
  Arms: Personal Resource Building and Inclusive Volunteering Intervention (PVI)
Other: Usual care — Usual stroke care services include medical and health services offered by the hospitals or community-based organisations.
  Arms: Control

SUMMARY:
This project will investigate effects of a novel theory-driven 6-week virtual Personal Resource Building and Inclusive Volunteering Intervention (PVI) on young stroke survivors' work ability, self-efficacy and psychosocial outcomes.

It is hypothesised that participants in the intervention group, compared with the control group, will demonstrate the outcomes below at immediately and 3 months post-intervention with respect to baseline: 1) Significant improvement in work ability (primary outcome), 2) Significant improvements in self-efficacy, health-related quality of life (HRQoL), emotional well-being and social skills (secondary outcomes).

Eligible participants will be randomly assigned to receive usual care or PVI with usual care and the control group participants will receive usual stroke care services.

DETAILED DESCRIPTION:
Returning to work is a major rehabilitation priority for young stroke survivors. This project will investigate effects of a novel theory-driven 6-week virtual Personal Resource Building and Inclusive Volunteering Intervention (PVI) on young stroke survivors' work ability, self-efficacy and psychosocial outcomes. A 2-arm, assessor-blind, randomised controlled trial will be conducted. Eligible participants will be randomly assigned to receive usual care or PVI with usual care and the control group participants will receive usual stroke care services. Outcomes including work ability, self-efficacy, health-related quality of life, emotional well-being and social skills will be measured at baseline, immediately post-PVI and 3 months post-PVI.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old,
* been clinically diagnosed with a first-ever or recurrent ischaemic or haemorrhagic stroke,
* living at home,
* Montreal Cognitive Assessment score >2nd percentile,
* a Modified Rankin Scale of 4 or below (moderately severe disability),
* able to communicate in Cantonese and read Traditional Chinese,
* a regular paid employment at the time of stroke,
* been unemployed for at least 3 months at the time of recruitment.

Exclusion Criteria:

* have been diagnosed with transient ischaemic attack,
* have experienced cerebrovascular events due to tumours,
* have been diagnosed with a mental condition such as depression, schizophrenia or bipolar disorder,
* demonstrate incomprehensible speech or difficulty in comprehending conversations, or
* have or are receiving vocational programmes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the level of perceived work ability | Change from baseline level to three months after completion of the intervention
  The Work Ability Index (Chinese version) will assess participants' perceived capability for work. It consists of 7 dimensions about participants' self-reported current work ability compared with the lifetime best. Total score is yielded by summing all items (range: 7-49): poor (7-27), moderate (28-36), good (37-43), and excellent (44-49) work ability.

SECONDARY OUTCOMES:
Change in the level of self-efficacy | Change from baseline level to three months after completion of the intervention
  The 10-item General Self-Efficacy Scale (GSES) (Chinese version) will assess participants' perceived self-efficacy in coping with stressful life events. Each item is rated on a 4-point scale (1=not at all true to 4=exactly true). Total score is yielded by summing all items (range: 10-40). A higher score indicates higher self-efficacy.
Change in the level of health-related quality of life | Change from baseline level to three months after completion of the intervention
  Participants' health-related quality of life (HRQoL) will be measured by the 47-item Stroke-Specific Quality of Life Scale (Chinese version). It has 11 domains on physical to psychosocial and participation. Items are scored from 1 (strongly disagree/cannot do it) to 5 (strongly agree/no trouble). Total score is yielded by summing all items (range 47-235). A higher score indicates higher HRQoL.
Change in the level of emotional well-being | Change from baseline level to three months after completion of the intervention
  The 14-item Hospital Anxiety and Depression Scale (HADS) (Chinese version) will measure participants' emotional well-being. Participants will rate their mood in the past week on a 4-point scale (0=no not at all to 3=yes definitely). It has 2 subscales (anxiety and depression). Subscale score is yielded by summing the relevant item scores (Total=0-21). A higher score indicates higher distress.
Change in the level of social skills | Change from baseline level to three months after completion of the intervention
  The 12-item Social Skills subscale of Work Personality Profile (Chinese version) will measure participants' interpersonal behaviours as applied to work. Item are rated on a 4-point scale (1=a problem area to 4=a definite strength). Total score is yielded by summing all items (range: 12-48). A higher score indicates greater proficiency in social skills at work.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Suzanne Lo, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The dataset will become available upon completion of the study upon written request made to the Principal Investigator.
Supporting Information: ICF
Time Frame: The data will become available upon completion of the study upon written request made to the Principal Investigator and for one year.
Access Criteria: The data will become available upon completion of the study upon written request made to the Principal Investigator.